CLINICAL TRIAL: NCT02693457
Title: Outcomes Following Suction Drain and Non-suction Drain Assisted Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Joint Replacement (Other)
Collaborators: University of Colorado, Denver (Other); CommonSpirit Health (Other)
Responsible Party: Principal Investigator, Jason Jennings, MD, Principal Investigator, Orthopedic Surgeon, Colorado Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1541
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis; Bilateral Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drain (Active Comparator): Intra-articular drain will be placed at closure of randomized knee for 24 hours
  Interventions: Procedure: Drain
- No Drain (Experimental): No intra-articular will be placed in the contralateral knee of the same patient. A placebo drain will be placed so patient is unaware of which knee contains working drain.
  Interventions: Procedure: No Drain

INTERVENTIONS:
Procedure: Drain — One randomized knee will be assigned to receive an intra-articular drain procedure following bilateral total knee arthroplasty. The drain will be removed 24 hours post-operatively. The patient will be blinded to fluid output from intra-articular drain.
  Arms: Drain
Procedure: No Drain — The contralateral knee will be assigned to a placebo drain procedure following bilateral total knee arthroplasty. This will blind the patient as to which knee contains the functioning intra-articular drain. A non-suction/ non-functional subcutaneous drain will act as the placebo drain. This drain will not output any fluid and will also be removed 24 hours after post-operatively.
  Arms: No Drain

SUMMARY:
This randomized controlled trial is designed to determine the effect of suction drain usage on the reduction of postoperative swelling following total knee replacement. Furthermore, this study will determine the relationship between postoperative swelling and quadriceps muscle function. This study will be performed in a cohort of patients undergoing bilateral total knee replacement and the suction intra-articular drain will be randomized to one of the two operative knees prior to surgery.

DETAILED DESCRIPTION:
This study has two primary aims: 1) to determine the effects of intra-articular suction drain use, placed during total knee arthroplasty (TKA), on postoperative knee joint effusion, which is the collection of fluid in the joint capsule, and lower extremity swelling compared to a TKA without the use of an intra-articular drain and, 2) to describe the relationship between postoperative lower extremity swelling and quadriceps function (strength and activation). The use of intra-articular drains during TKA surgery has been highly disputed, due to the fear of increasing risk of infection from a secondary incision site, however, past studies have found no increased risk of complication from drain use. Furthermore, studies have shown that drain use may reduce the amount of hidden blood loss, or blood that is collected in the intra-articular space. Of interest, effusion may be associated with decreased quadriceps function. Previous research examining the influence of knee effusion on quadriceps function has shown that with laboratory-induced acute knee effusion, quadriceps activation and force production are reduced. However, previous findings lack the ability to inform care for patients following TKA due to the acute nature of the effusion and the inability to translate findings from healthy individuals to a clinical population. This study has the potential to greatly improve care for patients undergoing TKA by informing the surgical procedure while also providing important evidence for the influence of postoperative swelling on quadriceps muscle function.

In order to maintain patient blinding, a non-functional subcutaneous drain will be placed in the non-randomized knee. Patients will be blinded to any fluid output from the intra-articular drain.

A medial parapatellar approach will be utilized for exposure of the knee. All TKAs will be performed using a gap balancing technique with substitution of the posterior collateral ligament (PCL). In all cases, a tensioning device will be used to establish balanced, symmetrical flexion and extension spaces. All TKA procedures will utilize cemented implants. Randomly assigned drains (intra-articular or subcutaneous) will be placed in respective knees before closure. All patients will be treated with Tranexamic Acid intravenously to standardize blood loss and effusion.

All patients will be provided standard rehabilitation protocol during their inpatient stay. After hospital discharge, patients will be encouraged to receive outpatient physical therapy 2-3 times per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 70 years
* Undergoing bilateral, simultaneous, primary knee replacements

Exclusion Criteria:

* neurological, vascular or cardiac problems that limit function
* unstable orthopedic conditions that limit functional performance
* previous history of inflammatory arthritis or other inflammatory systemic conditions
* previous history of deep vein thrombosis in either lower extremity
* lymphedema or other conditions that lead to lower extremity edema that may influence the outcomes of the study.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Isomechanical Dynomometery | 2 Weeks Post-Operative
  Knee Extensor Strength

SECONDARY OUTCOMES:
Lower Extremity Isomechanical Dynomometery | Pre-Operative
  Knee Extensor strength
Lower Extremity Hand Held Dyanmometry | 48 hours Post-Operative
  Knee Extensor strength
Lower Extremity Isomechanical Dynomometery | 6 Weeks Post-Operative
  Knee Extensor strength
Lower Extremity Isomechanical Dynomometery | 3 Month Post-Operative
  Knee Extensor strength
Clinical Quadriceps Activation Battery | Pre-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 8 hours Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 24 hours Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 48 Hours Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 2 weeks Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 6 weeks Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Clinical Quadriceps Activation Battery | 3 Months Post-Operative
  Isometric Quadriceps Set, Knee Extension Lag Test, Straight Leg Raise- Scale 0-6 (2 points for each test)
Bioelectrical Impedance for Swelling | Pre-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 8 hours Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 24 hours Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 48 Hours Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 2 Weeks Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 6 Weeks Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Bioelectrical Impedance for Swelling | 3 Months Post-Operative
  Using an RJL Systems Quantum Bioelectrical Impedance device, 4 electrodes will be placed on the subject's lower extremity (2 on calculated area of dorsum of foot, 2 on calculated area of anterior surface of thigh). A 425 microamp current at frequency 50kHz will be delivered to 2 electrodes. The remaining 2 electrodes will measure the voltage drop (in ohms) based on the resistance from body water content (swelling)
Circumferential Measure of Swelling | Pre-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 8 hours Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 24 hours Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 48 Hours Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 2 Weeks Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 6 Weeks Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Circumferential Measure of Swelling | 3 Months Post-Operative
  Using weighted, locking measuring tape, girth measurements will be taken at superior patellar pole and 10 cm proximal from superior patellar pole
Diagnostic Ultrasound Measure of Effusion | Pre-Operative
  Trained ultrasonagrapher will quantify the depth of effusion by summing the mm of effusion at three primary recesses (suprapatellar, medial parapatellar, lateral parapatellar). Diagnotic ultrasound will be performed with subject supine and knee flexed 30 degrees
Diagnostic Ultrasound Measure of Effusion | 48 Hours Post-Operative
  Trained ultrasonagrapher will quantify the depth of effusion by summing the mm of effusion at three primary recesses (suprapatellar, medial parapatellar, lateral parapatellar). Diagnotic ultrasound will be performed with subject supine and knee flexed 30 degrees
Diagnostic Ultrasound Measure of Effusion | 2 Weeks Post-Operative
  Trained ultrasonagrapher will quantify the depth of effusion by summing the mm of effusion at three primary recesses (suprapatellar, medial parapatellar, lateral parapatellar). Diagnotic ultrasound will be performed with subject supine and knee flexed 30 degrees
Diagnostic Ultrasound Measure of Effusion | 6 Weeks Post-Operative
  Trained ultrasonagrapher will quantify the depth of effusion by summing the mm of effusion at three primary recesses (suprapatellar, medial parapatellar, lateral parapatellar). Diagnotic ultrasound will be performed with subject supine and knee flexed 30 degrees
Diagnostic Ultrasound Measure of Effusion | 3 Months Post-Operative
  Trained ultrasonagrapher will quantify the depth of effusion by summing the mm of effusion at three primary recesses (suprapatellar, medial parapatellar, lateral parapatellar). Diagnotic ultrasound will be performed with subject supine and knee flexed 30 degrees
Knee Pain Measured by Visual Analog Scale | Pre-Operative
Knee Pain Measured by Visual Analog Scale | 8 Hours Post-Operative
Knee Pain Measured by Visual Analog Scale | 24 Hours Post-Operative
Knee Pain Measured by Visual Analog Scale | 48 Hours Post-Operative
Knee Pain Measured by Visual Analog Scale | 2 Weeks Post-Operative
Knee Pain Measured by Visual Analog Scale | 6 Weeks Post-Operative
Knee Pain Measured by Visual Analog Scale | 3 Months Post-Operative
Knee Flexion Range of Motion | Pre-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 8 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 24 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 48 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 2 Weeks Post Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 6 Weeks Post Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Flexion Range of Motion | 3 Months Post Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | Pre-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 8 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 24 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 48 Hours Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 2 Weeks Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 6 Weeks Post-Operative
  Active and Passive Range of Motion Measured with Goniometer
Knee Extension Range of Motion | 3 Months Post-Operative
  Active and Passive Range of Motion Measured with Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

REFERENCES:
- [Background] Esler CN, Blakeway C, Fiddian NJ. The use of a closed-suction drain in total knee arthroplasty. A prospective, randomised study. J Bone Joint Surg Br. 2003 Mar;85(2):215-7. doi: 10.1302/0301-620x.85b2.13357. PMID 12678355
- [Background] Holt BT, Parks NL, Engh GA, Lawrence JM. Comparison of closed-suction drainage and no drainage after primary total knee arthroplasty. Orthopedics. 1997 Dec;20(12):1121-4; discussion 1124-5. doi: 10.3928/0147-7447-19971201-05. PMID 9415907
- [Background] Palmieri-Smith RM, Villwock M, Downie B, Hecht G, Zernicke R. Pain and effusion and quadriceps activation and strength. J Athl Train. 2013 Mar-Apr;48(2):186-91. doi: 10.4085/1062-6050-48.2.10. Epub 2013 Feb 20. PMID 23672382
- [Background] Pietrosimone B, Lepley AS, Murray AM, Thomas AC, Bahhur NO, Schwartz TA. Changes in voluntary quadriceps activation predict changes in muscle strength and gait biomechanics following knee joint effusion. Clin Biomech (Bristol). 2014 Sep;29(8):923-9. doi: 10.1016/j.clinbiomech.2014.06.014. Epub 2014 Jul 4. PMID 25062605